CLINICAL TRIAL: NCT04508764
Title: Implementation of the Families Accelerating Cascade Testing Toolkit (FACTT) for Hereditary Breast and Ovarian Cancer and Lynch Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding and slow enrollment
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 202006168
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Hereditary Breast and Ovarian Cancer; Lynch Syndrome
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): * For approximately the first 6 months of the study, or until 75 patient with cancer who is initially approached in clinic (probands) are enrolled, the investigators will be enrolling probands into the "Usual Care" group. During this time, the investigators will clarify usual care regarding cascade genetic testing for each participating clinic and proband participant. The investigators will do this by proband participant surveys, as well as initial provider semi-structured interviews.
  * Proband: Complete Cascade Genetic Testing survey. The survey will also contain questions regarding willingness or not to invite each eligible 1st degree family member to participate in the family study. At 6 months, there will be a follow-up survey
  * Family Member: Complete survey at study entry and at 6 month follow-up
- FACT Toolkit (FACTT) (Experimental): * Proband: Introduced to FACTT and will complete Cascade Genetic Testing survey. The survey will contain questions regarding willingness or not to invite each eligible 1st degree family member to participate in the family study. The probands will also fill out assessments of each FACTT component. At 6 months, there will be a follow-up survey.
  * Family Member: Introduced to FACTT and will complete surveys at study entry and 6 month follow-up. They will also fill out assessments of each FACTT component
  Interventions: Other: Families Accelerating Cascade Testing Toolkit

INTERVENTIONS:
Other: Families Accelerating Cascade Testing Toolkit — -Online family history assessment, video of Siteman Cancer Center genetic counselors, physicians and patients highlighting the importance of cascade genetic testing, reviewing and receiving a family letter and gene information sheet, reviewing websites/online resources, and offering a family visit with a genetic counselor
  Other Names: FACTT
  Arms: FACT Toolkit (FACTT)

SUMMARY:
The purpose of this research study is to learn how cancer care providers can help their patients communicate the need for genetic testing in families with inherited cancer syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of HBOC or Lynch-associated "pathogenic/ likely pathogenic" mutation per American College of Medical Genetics and Genomics criteria (1)
* Diagnosis of one or more invasive cancers: epithelial ovarian, fallopian tube, primary peritoneal, breast, colorectal, endometrial
* Mutation listed in NCCN guidelines with at least Category 2A evidence for intervention
* Over the age of 18
* Psychological ability and general health that permits completion of study requirements and follow-up
* Willingness to complete follow-up surveys in person, electronically, or by telephone for up to 6 months

Exclusion Criteria:

-"Variant of undetermined significance," "likely benign" or "benign" variant per ACMGG criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Proband-reported cascade testing rates of first-degree relatives | From start of study through completion of 6 month follow-up (estimated to be 18 months)
  -For each proband, this testing rate is defined as the number of first-degree relatives tested divided by the number of living first-degree relatives age-appropriate for testing, as determined by family surveys done by the proband. The investigators will calculate mean cascade genetic testing rates for both conditions (Usual Care and FACTT intervention).
Number of primary barriers to genetic testing for first-degree relatives | From start of study through completion of 6 month follow-up (estimated to be 18 months)
  -The Cascade Genetic Testing survey will assess knowledge, perception, and personal experience with sharing germline mutation information with first-degree relatives
Family member-reported cascade testing rates | From start of study through completion of 6 month follow-up (estimated to be 18 months)
  -This testing rate is defined by the number of family members tested divided by the number of living family members age-appropriate for testing
Number of primary barriers to genetic testing for family members | From start of study through completion of 6 month follow-up (estimated to be 18 months)
  -The Family Member survey will assess experience with considering testing themselves, decisional regret regarding genetic testing, and if they have tested positive

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Hagemann, M.D., MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu